CLINICAL TRIAL: NCT02935699
Title: A Phase III, Multi-center, Double Blind, Randomized, Active Controlled Clinical Trial to Evaluate the Non-Inferiority Comparing Cetirizine Injection 10 mg to Diphenhydramine Injection, 50 mg, for the Treatment of Acute Urticaria
Brief Title: Clinical Trial Comparing JDP-205 to Diphenhydramine Injection for the Treatment of Acute Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JDP Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETTAU-03
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Acute Urticaria
MeSH Terms: interventions — Drug Evaluation; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): JDP-205 Injection, 10 mg/mL, 1 mL
  Interventions: Drug: Test Drug (JDP-205)
- Control (Active Comparator): Diphenhydramine Injection, 50 mg/mL, 1 mL
  Interventions: Drug: Active Control (Diphenhydramine)

INTERVENTIONS:
Drug: Test Drug (JDP-205) — Cetirizine, 10mg/mL; a single 1.0 mL injection via intravenous (IV) push over a period of ~2 minutes
  Other Names: QUZYTTIR
  Arms: Test Drug
Drug: Active Control (Diphenhydramine) — Diphenhydramine Injection, 50 mg/mL;a single 1.0 mL injection via intravenous (IV) push over a period of ~2 minutes
  Other Names: Benadryl
  Arms: Control

SUMMARY:
This is a multicenter, parallel group, randomized, double-blind, active controlled, Phase III clinical study of cetirizine injection, 10 mg/mL, compared to diphenhydramine injection, 50 mg/mL (Benadryl or generic equivalent) with acute urticaria requiring treatment.

DETAILED DESCRIPTION:
This was a multi-center, parallel group, randomized, double-blind, active controlled, Phase III clinical trial of cetirizine injection 10 mg/mL versus diphenhydramine injection 50 mg/mL (Benadryl or generic equivalent) in approximately 256 subjects who either presented to Emergency Departments, hospitals, allergy clinics or Urgent Care Centers with acute urticaria, or developed acute urticaria following allergen challenge at an Allergy Clinic.

Patients signed an informed consent and were evaluated for eligibility for inclusion to treat. Eligible subjects were assessed for baseline characteristics, medical and surgical histories, concomitant medications and given a brief physical exam.

Subjects were then randomized, in a 1:1 ratio, to blindly receive either cetirizine 10 mg/mL injection or diphenhydramine 50 mg/mL injection.

Efficacy assessments included patient-rated severity of pruritus, physician assessments of extent of urticaria/erythema, and sedation score. Subjects remained in the treatment center for at least after the 1 hr assessment, after which they may have been discharged at the physician's discretion.

Safety was monitored through the reporting of adverse events for up to 28 days following treatments and by monitoring vital signs at planned intervals from admission into the treating facility until readiness for discharge. After 24 and 48 hrs after discharge, subjects were contacted by phone for follow-up questions regarding recurrence of symptoms, new symptoms, additional medication taken, side effects from medication taken after discharge, relapse requiring a return to treatment center, and return to normal activities.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with a diagnosis of acute urticaria who need treatment with antihistamine to alleviate their symptoms;
2. 18 years of age or older;
3. Be willing and able to give informed consent;
4. Patients with a Patient rated Pruritus Severity Score ≥ 1

Exclusion Criteria:

1. Receipt of an investigational drug or device, within the past 30 days;
2. Patients in whom an antihistamine may be contraindicated (e.g. narrow angle glaucoma, symptomatic prostatic hypertrophy);
3. Patients who, in the opinion of the investigator, may not tolerate an IV injection of diphenhydramine 50 mg, or cetirizine 10 mg;
4. Receipt of any antihistamine (H1 antagonist) within the past 2 hours regardless of the route of administration, e.g. diphenhydramine, cetirizine, loratadine, fexofenadine, levocetirizine, desloratadine;
5. Receipt of an H2 antagonist within the past 2 hours;
6. Receipt of doxepin within the past 2 hours; doxepin is an antidepressant, but it also has antihistamine properties;
7. Receipt of steroids by the oral, IV, IM, or inhalational routes route within the past 4 hours to manage an acute allergic reaction;
8. Receipt of epinephrine (EpiPen or any other brand) within the past 20 minutes;
9. Anaphylaxis prior to the acute anaphylactic symptoms having been treated.
10. Has known allergy to hydroxyzine, cetirizine or levocetirizine, or diphenhydramine;
11. Pregnancy or breastfeeding;
12. Patients who have an acute allergic reaction to medication they are taking (e.g. antibiotics, NSAIDs, etc.) and who cannot stop the medication;
13. Patients who, based on their medical history or in the opinion of the investigator, have chronic urticaria, hereditary angioedema, urticaria refractory to antihistamines, or dermatological disease that interferes with evaluation of a therapeutic response;
14. Any condition that in the view of the investigator makes the subject unsuitable for enrollment in this study;
15. History of HIV or other known immunodeficiency;
16. Major medical or psychiatric illness, other than acute urticaria, at the time of presentation;
17. Inability to provide informed consent.
18. Patients on concomitant p-glycoprotein inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JIE DU, PH.D., Study Chair — JDP Therapeutics, Inc.
Locations (4):
- United States (3):
  - Univ of Cincinnati Medical Center, Cincinnati, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - City Doc Urgent Care center, Dallas, Texas
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abella BS, Berger WE, Blaiss MS, Stiell IG, Herres JP, Moellman JJ, Suner S, Kessler A, Klausner HA, Caterino JM, Du J. Intravenous Cetirizine Versus Intravenous Diphenhydramine for the Treatment of Acute Urticaria: A Phase III Randomized Controlled Noninferiority Trial. Ann Emerg Med. 2020 Oct;76(4):489-500. doi: 10.1016/j.annemergmed.2020.05.025. Epub 2020 Jul 9. PMID 32653333
- See also: Sponsor website — http://jdptherapeutics.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Drug: JDP-205 Injection, 10 mg/mL, 1 mL
  Test Drug (JDP-205): JDP-205 Injection, 10 mg/mL, 1 mL
- Control: Diphenhydramine Injection, 50 mg/mL, 1 mL
  Active Control (Diphenhydramine): Diphenhydramine Injection, 50 mg/mL
Period: Overall Study
Arm/Group | Test Drug | Control
Started | 127 | 135
Completed | 127 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Drug | Control | Total
Number analyzed (Participants) | 127 | 135 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (16.28) | 39.2 (15.96) | 39.1 (16.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 88 | 165
  Male | 50 | 47 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 41 | 44 | 85
  White | 64 | 62 | 126
  More than one race | 17 | 24 | 41
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 135 | 262

OUTCOME MEASURES:

1. Primary Outcome: Change of Patient Rated Pruritus Score
Description: Change from baseline to 2 hours in patient-rated pruritus Severity score (values at 2 hours minus Baseline)
  Patient Pruritus Severity Score Ask the patient "How severely are your hives itching at the moment?" 0 = none
  1. = mild (minimal awareness, easily tolerated)
  2. = moderate (definite awareness, quite bothersome)
  3. = severe (difficult to tolerate)
Time Frame: 2 hr
Population: Intent To Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 127 | 135
score on a scale | -1.61 (0.944) | -1.50 (0.984)

2. Secondary Outcome: Number of Patients Who Needed to Return to Treatment Center
Description: Number of patients who needed to return to treatment center approximately 24 hours after discharge
Time Frame: up to 24 hrs
Population: Intent To Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 127 | 135
Participants | 7 | 19

3. Secondary Outcome: Time to Discharge
Description: Time spent (hours) at the treatment center
Time Frame: up to 24 hours
Population: Intent To Treat Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 127 | 135
hours | 1.71 (0.868) | 2.07 (1.112)

4. Secondary Outcome: Patient Sedation Scores
Description: Patient Sedation Score at 2 hours
  Ask the patient "How drowsy do you feel at the moment?" 0 = None (Not drowsy at all)
  1. = Mild (Slightly drowsy)
  2. = Moderate (Quite drowsy)
  3. = Severe (Extremely drowsy)
Time Frame: 2 hours
Population: Intent To Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 127 | 135
score on a scale | 0.46 (0.721) | 0.88 (0.955)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Test Drug | Control
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/127 | 1/135
Other Adverse Events (participants affected / at risk) | 5/127 | 18/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Drug (N=127) | Control (N=135)
anaphylactic reaction (Immune system disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Drug (N=127) | Control (N=135)
Dizziness (Nervous system disorders) | 0 | 6
Burning sensation (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (Injury, poisoning and procedural complications) | 0 | 2
Feeling hot (Injury, poisoning and procedural complications) | 1 | 0
Injection site pain (Injury, poisoning and procedural complications) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT02935699/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT02935699/SAP_001.pdf